CLINICAL TRIAL: NCT02950493
Title: Use of Reactivated DEFINITY or Lumason in Patients Undergoing Rest or Stress Echocardiography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In none of the patients could acoustic activation be produced
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0281-16-FB
Record Dates: First submitted 2016-09-14; First posted 2016-11-01 (Estimated); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Stress Echocardiography
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single group, one arm study group (Other): Compare echocardiograph imaging efficacy of active Definity or Lumason (perflutren lipid microsphere) with compressed Definity or Lumason.
  Interventions: Other: perflutren lipid microsphere

INTERVENTIONS:
Other: perflutren lipid microsphere — Definity and Lumason are tools for diagnosis used in echocardiography. Compare activated Definity or Lumason with compressed Definity or Lumason.
  Other Names: DEFINITY; LUMASON

SUMMARY:
Use of Reactivated DEFINITY® in or LUMASON Patients Undergoing Rest or Stress Echo Purpose of the study: Each patient undergoing a rest or stress echocardiogram uses a full vial of DEFINITY® or LUMASON contrast agent. During infusion, this often condenses back to its liquid phase due to manual pressure applied in the syringe. At this point, it is not optimal to be used at current ultrasound settings for stress echocardiography. This research project will test whether this condensed DEFINITY® or LUMASON can be reactivated by ultrasound using the same transducer used to image the patient.

Eligibility: Same criteria as required for stress echo procedure. Interventions and Evaluations: Inject condensed DEFINITY® or LUMASON at end of stress test Follow Up: The patient would be observed by echo lab staff for half an hour following completion of the stress test. There would be no longitudinal follow up.

DETAILED DESCRIPTION:
Patients undergoing previously scheduled rest or stress echocardiography with the primary investigator as the supervising physician will be identified and consented. The standard stress echocardiography procedure will be performed. Definity® or LUMASON will be removed from refrigeration and agitated for 45 seconds to vaporize into its gaseous phase. One mL of Definity® or LUMASON will then be diluted in 29 mL of isotonic, sterile saline. Patients will undergo baseline echocardiography followed by stress with either dobutamine or exercise. Standard Definity® or LUMASON will be injected intravenously into the subject via peripheral intravenous access obtained prior to the study by a registered nurse at the end of the rest or stress portion of the procedure coinciding with image acquisition. Contrast enhanced echocardiography by standard acoustic acquisition will be performed following rest or stress for the indicated diagnostic purpose of the test. By the end of the exam, the gaseous Definity® or LUMASON will have undergone manual compression via manual pressure and condensed back to its liquid phase. At this point, the compressed Definity® or LUMASON will be given intravenously with repeated transthoracic echocardiography. During this second round of image acquisition, real time (RT) imaging (35 Hertz) and 1:1 triggered (Tr) end systolic imaging at various mechanical indices (MI's) up to 1.2 will be performed in standard transthoracic echocardiography windows. Acoustic Intensity (AI) within the left ventricular (LV) cavity, the anterior myocardium (AM) and inferolateral myocardium (ILM) at end systole will be obtained at each MI setting with real time or triggered imaging. Differences in AI between Tr and RT imaging within the AM and ILM at each MI will be used to quantify bubble activation/destruction. Following image acquisition, the patient will be observed for 30 minutes by echo lab staff with nearby resuscitative equipment per current protocol. If no adverse events are noted, the patient will then be dismissed.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older at screening
* Clinically indicated stress echocardiography to take place at the UNMC echocardiography laboratory

Exclusion Criteria:

* Prior allergic reaction to Definity® or Lumason
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Acoustic index | Data obtained at time of stress echo and all data will be acquired and study completed within 1 hour of stress echo or regular echo study. No follow up is needed or indicated.
  Acoustic index during realtime and triggered imaging between compressed Definity or Lumason and activated Definity or Lumason

SECONDARY OUTCOMES:
Clinical Adverse Events regarding reading of echocardiography | The data will be obtained within 30 minutes of the echocardiogram or stress echocardiogram. Any potential side effects will have occurred within this time frame as well.
  Monitor for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data.